CLINICAL TRIAL: NCT04712929
Title: Association of Candida and Antifungal Therapy With Pro-inflammatory Cytokines in Oral Leukoplakia- A Pilot Study
Brief Title: Candida Associated Cytokines in Oral Leukoplakia
Status: Completed | Type: Observational
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Dr. Shalini Gupta, Associate Professor, All India Institute of Medical Sciences
Other Study IDs: A-634
Record Dates: First submitted 2021-01-11; First posted 2021-01-19 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Oral Leukoplakia
Keywords: Candida; oral leukoplakia; il 6; il 8; il 17; TNF alpha; aspartyl proteinase; biofilm formation; phospholipase; antifungal sensitivity
MeSH Terms: conditions — Leukoplakia, Oral; Torulopsis | interventions — Fluconazole; Behavior Therapy; Tobacco Products; Catechin; Ethanol

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Homogenous oral leukoplakia: uniform, flat, thin, smooth/ wrinkled/corrugated surface throughout the white lesion.
  Tab Fluconazole 100 mg as a mouthwash ( tablet dissolved in 10 ml of drinking water and used as a mouth rinse for 2 minute and swallowed) once a day for 14 days
  Interventions: Other: Fluconazole
- Non-Homogenous oral leukoplakia: mixture of red and white lesions with a irregularly speckled/ nodular/ verrucous surface Tab Fluconazole 100 mg as a mouthwash ( tablet dissolved in 10 ml of drinking water and used as a mouth rinse for 2 minute and swallowed) once a day for 14 days
  Interventions: Other: Fluconazole
- Control group: 30 healthy controls ( age and sex matched) would also be recruited from patients who are reporting for other routine dental problems.

INTERVENTIONS:
Other: Fluconazole — ( Tab Fluconazole 100 mg as a mouthwash ( tablet dissolved in 10 ml of drinking water and used as a rinse for 2 minute and swallowed) once a day for 14 days WHO criteria 5As and 5Rs for tobacco cessation
  Other Names: Behavioral intervention for tobacco/ betel nut / alcohol cessation
  Groups: Homogenous oral leukoplakia; Non-Homogenous oral leukoplakia

SUMMARY:
This study aims to determine the correlation between candida and pro- inflammatory cytokines response in Oral Leukoplakia(OL) with antifungal therapy. Ethical clearance from the Institutes ethical committee and Informed written consent from the patient will be obtained. The study group would comprise of clinically and histopathologically confirmed cases of OL (60 patients). The control group would be 30 dental patients ( age & sex matched) who do not any malignancy, OL or any other potentially malignant disorder of oral mucosa. Patients who have any predisposing factor for oral candidiasis will be excluded from the study. Swabs will be taken from the oral lesion and cultured for candida to determine phenotypes, virulence attributes and antifungal sensitivity. Sterile PVA opthalmic sponges will be used to collect sample from the surface of oral epithelium and then processed to determine levels of pro- inflammatory cytokines (IL-6, IL-8. IL-17, TNFα). This procedure will be repeated in study group 2 weeks after a course of antifungal therapy. The results will be tested statistically at a confidence level of 95%.

DETAILED DESCRIPTION:
Objectives

1. To determine the association of candida phenotypes, virulence attributes ( Secreted aspartyl proteinases, biofilm formation, Phospholipase) and antifungal sensitivity with clinicopathologic characteristics in oral leukoplakia
2. To determine the secretion and levels of pro-inflammatory cytokines ( IL-6, IL-8. IL-17, TNFα ) in oral leukoplakia before and after antifungal therapy.
3. To study the correlation between candida and pro-inflammatory cytokines in oral leukoplakia with antifungal therapy

Detailed methodology including study design, outcome measures, sample size and statistical analysis.

Study design:

Prospective case- control observational study

Selection of patients:

The patients in the study group and control group will be consecutively recruited from the Oral Medicine & Radiology clinic at Centre for Dental Education & Research AIIMS.

Sample size:

The study will include 60 OL ( 30 Homogenous OL, 30 Non- Homogenous OL) and 30 healthy controls

Clinicopathologic characteristics:

The clinical characteristics and staging/grading would be recorded as per prepared proforma for each group. Written informed consent would be taken before any further investigation. History of tobacco, betel nut, alcohol habits with frequency, duration of habit and current status, oral burning sensation with Visual Analogue Scale (VAS) scores will be Routine blood investigations would be done before incisional biopsy and histopathological confirmation of the diagnosis. The H & E histopathological features with Periodic Acid Schiff (PAS) staining would be recorded and grading done for study group as per standard World Health Organization criteria. The clinical staging of OL will be done as per OL staging system (OLEP) ( van der Waal 2000) with photographic records of lesions by two calibrated observers.Tobacco,betel nut and alcohol cessation counselling and oral hygiene instructions will be given.

Sample collection for study:

A). Candida phenotypes, virulence and antifungal sensitivity study. Collection , transport and processing: Two oral swabs from each patient ( pre-wet with sterile normal saline) will be taken from the oral lesion and sent to the Mycology Laboratory, Department of Microbiology for further processing as per standard laboratory procedures.

Direct microscopy: One swab sample will be examined by microscopy for detection of yeast cells by preparing gram stain.

Culture: The second swab will be inoculated on Sabouraud dextrose agar (SDA) medium with gentamicin and will be kept at 37°C for incubation for 48 hours. Gram staining will be performed on any growth morphologically resembling to that of yeast.

Phenotypic identification: Identification of isolates was performed by using germ tube, morphology on corn meal agar, colour on triphenyl tetrazolium chloride and CHROM agar medium Determination of virulence factors of Candida spp Various virulence factors like phospholipase activity, Secreted aspartyl proteinase (SAP) and Biofilm formation (BF) will be determined as per the standard protocol.

Determination of Phospholipase (PL) activity Phospholipase activity will be measure by growing cells on egg yolk agar medium and measuring the size of the zone of precipitation. A cell suspension of 106 yeast cells/ml in saline will be prepare and 5μl will be place on the surface of the egg yolk medium. The culture will then incubated at 37°C for 7-8 days, after which the diameter of the precipitation zone around the colony will be determine. Phospholipase activity (Pz) will be measure by dividing colony diameter by the diameter of the precipitation zone (pz) around the colony formed on the plate. Each isolate will be tested in duplicate. The C. albicans SC 5314 strain will be used as positive control.

Determination of Secreted aspartyl proteinase (SAP) activity All isolates will be tested for their ability to grow and produce a clear zone of hydrolysis in bovine serum albumin (BSA) agar. . A 5μl of 1x106 cells /ml will be placed on solid medium and will be incubated at 37°C for 3-4 days. Subsequently, clearing of the opacity by hydrolysis of precipitated albumin will be recorded. The C. albicans SC 5314 strain will be used as positive control.

Determination of Biofilm formation (BF) A 100μl volume of 1 x 106 cells /ml suspension will be place on sterile, polystyrene, flat-bottom 96-well microtitre plates and will be incubated for 48 h at 37°C for adherence and biofilm. After 48 hr wells will be washed with PBS and a semi-qualitative measure of biofilm will be detected by XTT [2,3-bis (2-methoxy-4nitro-5-sulfo-phenyl) - 2H - tetra-zolium-5-carboxanilide] -reduction assay A colorimetric change in the XTT-reduction assay, a direct correlation of the metabolic activity of the biofilm, will then be measure in a microtiter plate reader at 490 nm after 2 hr of incubation.

Antifungal susceptibility testing of isolates Antifungal susceptibility for voriconazole fluconazole and clotrimazole will be performed by disk diffusion method as per the CLSI M44-A2 recommendation on the yeast isolates.

B). Pro- Inflammatory cytokines study Sample collection of oral secretions from lesion Four Sterile PVA ophthalmic sponges (Merocel) will be used to collect samples of oral secretions for four pro-inflammatory cytokine study from the oral lesion (other than biopsy site). This is a non- invasive method and makes it site -specific which is an advantage over other serum and saliva estimations. In addition, assessment of local cytokine levels via longitudinal sampling in patients undergoing antifungal therapy in OL may allow for an understanding of the temporal nature of cytokine elevation and clinical response to antifungals.

This procedure will be done for both the study group and control group. The subjects will be asked to abstain from eating, drinking and rinsing the mouth at least 2 hours prior to sampling. The sponges will be pre-wet with sterile normal saline, kept in contact with the lesion without rubbing or movement or 1 minute and then immediately stored in sterile containers at -80 °C till further analysis in Biochemistry department AIIMS. A photographic and clinical record of the sample site will be kept with the patient proforma for future reference. This procedure will be repeated at the same site after antifungal therapy for study group and a photographic record will be kept for comparison. Ethical clearance from Institute ethics board will be taken. Informed written consent will be obtained and information regarding the study would be given to the study subjects and controls prior sample collection.

Estimation of IL-6, IL-8, IL-17 and TNFα levels by ELISA The opthalmic sponges (Merocel ) will be thawed at room temperature for 10 min. Sponges will then be inserted into a microcentrifuge tube containing a 0.2 μm filter (SpinX centrifuge tube), equilibrated by adding 300 μl of extraction buffer and incubated for 30 min at 4 °C, followed by centrifugation at 4 °C for 30 min at 14,000 rpm. After centrifugation, the resultant supernatant will be collected for the estimation of IL-6, IL-8, IL-17 and TNFα levels by ELISA method with commercially available kits. The supernatant will be stored at -80 °C until use.

A monoclonal antibody against the antigens (IL-6, IL-8, IL-17 and TNFα) has been pre-coated onto the wells of the microtiter strips provided. Antigens present in the sample or standard will be incubated with the plates to allow binding of antigens to the antibody. This is followed by the addition of a primary monoclonal anti- IL-6, IL-8, IL-17 and TNFα antibody respectively conjugated to biotin in respective microtiter plates. An avidin-HRP conjugated antibody specific for primary antibody will then be added to the wells. After incubation and following a wash, to remove any unbound antibody enzyme reagent, a TMB one-step substrate reagent reactive with HRP will be added to the wells. The color development will be terminated by adding acid and absorbance was measured at 450 nm. A reference curve will be obtained by plotting the different concentrations of standard samples versus absorbance and levels of the antigens in samples tested will be calculated by its standard plot.

Antifungal therapy The study group will be treated with antifungal therapy ( Tab Fluconazole 100 mg as a mouthwash ( tablet dissolved in 10 ml of drinking water and used as a rinse for 2 minute and swallowed) once a day for 14 days). The procedure will be demonstrated to each study subject before starting the treatment. The oral burning sensation and clinical characteristics of the lesions with intraoral photographs will be recorded after antifungal therapy.

Statistical analysis:

The distribution of candida phenotypes, virulence attributes and antifungal sensitivity in the study and control groups would be correlated with levels of IL-6, IL-8, IL-17 and TNFα and clinicopathological characteristics. Correlations between virulence factors and clinical characteristics will be determined. Cohens kappa statistic will be used to determine intraobserver reliability. A comparison of the levels of pro inflammatory cytokines(IL-6, IL-8, IL-17 and TNFα) before and after antifungal therapy will be done in the study group. The results would be tested for statistical significance.The Chi- square and the Mann- Whitney U tests will be used to estimate the statistical significance of difference observed between the groups.

7.Ethical Clearance Obtained

ELIGIBILITY:
Inclusion criteria:

* 60 clinically and histologically confirmed cases of Oral Leukoplakia would be prospectively recruited for this study who have not been under treatment for the same for past 6 months.
* 30 healthy controls ( age and sex matched) would also be recruited from patients who are reporting for other routine dental problems.
* Also these patients would be those who have good oral hygiene (simplified oral hygiene index score 0-3, periodontal screening and recording PSR code 0-2) and do not have any potentially malignant disorder of the oral mucosa or oral squamous cell carcinoma and have no systemic diseases or any other malignancy.

Exclusion criteria:

* Patients with history of significant and serious uncontrolled systemic disease allergy to antifungals or history of antifungal therapy in past 6 months.
* Patients with history of any other malignant disease.
* Children ( age < 18 years) and pregnant women.
* Patients with history of major/ minor surgery and predisposing factors for oral candidal infection like diabetes/ endocrine disorders, xerostomia, poor oral hygiene, removable prosthesis, prolonged corticosteroid/ antibiotic/ immunosuppressant/ antibacterial mouthwash therapy, radiation/ chemotherapy, auto immune disorders and primary / secondary immune deficiencies, nutritional deficiencies and hospitalized debilitated patients.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patients in the study group and control group will be consecutively recruited from the Oral Medicine & Radiology clinic at Centre for Dental Education & Research AIIMS.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-02-15 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Oral burning sensation | Before and after antifungal treatment (2 weeks)
  VAS score (0-10)
Clinical size of lesion | Before and after antifungal treatment (2 weeks)
  maximum Length( L) and width (W) L1: L/W ≤ 2 cm L2: L /W 2-4 cm L3: L/W ≥ 4cm
Pro- inflammatory cytokines | Before and after antifungal treatment (2 weeks)
  il6,il8,il17,TNF-alpha by ELISA before and after antifungal treatment
Erythema of oral lesion | Before and after antifungal treatment (2 weeks)
  Scores as [ 0- no change, 1- minimal change ( Reduction in erythema < 1cm of oral lesion, and 2- significant change( Reduction in erythema ≥ 1cm of oral lesion)
Thickness of oral lesion | Before and after antifungal treatment (2 weeks)
  Scores as [ 0- no change, 1- minimal change ( Reduction in thickness < 1cm of oral lesion, and 2- significant change( Reduction in thickness ≥ 1cm of oral lesion)
candida positivity | before antifungal treatment
  Swabs for smear or culture positive for Candida
Phospholipase Activity of Candida in Oral leukoplakia | Before antifungal therapy
  Phospholipase activity (Pz) was measured by dividing colony diameter by the diameter of the precipitation zone (Pz) around the colony formed on the plate. A Precipitation zone (in mm) around colony 1.0 : 0 negative (-), 0.99-0.9 : 1 weak (+), 0.89-0.8: 2 poor (++), 0.79-0.7: 3 moderate (+++), < 0.69: 4 Strong positive(++++),
Secreted aspartyl proteinase activity of Candidain Oral leukoplakia | Before antifungal therapy
  Secreted aspartyl proteinase activity was measured by dividing colony diameter by the diameter of the precipitation zone (Pz) around the colony formed on the plate. A Precipitation zone (in mm) around colony 1.0 : 0 negative (-), 0.99-0.9 : 1 weak (+), 0.89-0.8: 2 poor (++), 0.79-0.7: 3 moderate (+++), < 0.69: 4 Strong positive(++++),
Biofilm formation | Before antifungal therapy
  Absorbance values of test wells at 490nm of XTT reduction assay- absorbance values of control
Antifungal sensitivity | Before antifungal therapy
  Using CLSI document M44-A for disk diffusion method for Fluconazole (25 μg), Voriconazole (1 μg) and Clotrimazole (50 μg) S: Sensitive R: Resistant I: Intermediate
Histopathology | Before antifungal therapy
  Mild Dysplasia Moderate Dysplasia Severe Dysplasia PAS stain positive/ negative

SECONDARY OUTCOMES:
Malignant transformation | after 2,5,7,10 years
  Histological features of Oral Squamous Cell Carcinoma

CONTACTS AND LOCATIONS:
Overall Officials: Shalini Gupta, MDS,FDSRCS, Principal Investigator — All India Institute of Medical Sciences
Locations (1):
- All india Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gupta SR, Gupta N, Sharma A, Xess I, Singh G, Mani K. The association of Candida and antifungal therapy with pro-inflammatory cytokines in oral leukoplakia. Clin Oral Investig. 2021 Nov;25(11):6287-6296. doi: 10.1007/s00784-021-03927-3. Epub 2021 Apr 4. PMID 33813637